CLINICAL TRIAL: NCT04180449
Title: DYsphagiA in interMedIate Care UnitS - a Retrospective Analysis of Available Data
Brief Title: DYsphagiA in interMedIate Care UnitS
Acronym: DYnAMICS II
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: DYnAMICS II
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagia screening positive
  Interventions: Other: Screening for dysphagia along clinical routine
- Dysphagia screening negative
  Interventions: Other: Screening for dysphagia along clinical routine

INTERVENTIONS:
Other: Screening for dysphagia along clinical routine — Screening for dysphagia using the water swallow test in intermediate care unit patients

SUMMARY:
Retrospective study in intermediate care unit patients on the incidence, Risk factors, and effects on mortality of dysphagia. During a 6-month observational period, routine data will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate care unit patients admitted within the observational period

Exclusion Criteria:

* documented refusal to General Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intermediate Care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of positive screening (first screening) for dysphagia in neurosurgical intermediate care unit patients | within 8 hours from intermediate care unit admission
  incidence: percentage of patients with screening positivity at first screening

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Intensive Care Medicine, Bern, Switzerland

REFERENCES:
- [Background] Zuercher P, Moret CS, Dziewas R, Schefold JC. Dysphagia in the intensive care unit: epidemiology, mechanisms, and clinical management. Crit Care. 2019 Mar 28;23(1):103. doi: 10.1186/s13054-019-2400-2. PMID 30922363
- [Background] Schefold JC, Berger D, Zurcher P, Lensch M, Perren A, Jakob SM, Parviainen I, Takala J. Dysphagia in Mechanically Ventilated ICU Patients (DYnAMICS): A Prospective Observational Trial. Crit Care Med. 2017 Dec;45(12):2061-2069. doi: 10.1097/CCM.0000000000002765. PMID 29023260